CLINICAL TRIAL: NCT06035445
Title: Interactive Transition Support for Adolescents Living With HIV Comparing Virtual and In-person Delivery Through a Stepped-wedge Cluster Randomized Clinical Trial in South Africa
Brief Title: Support for Adolescents Living With HIV in South Africa
Acronym: InTSHA VIP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: University of KwaZulu (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Brian Zanoni, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00004803; 1R01MH131434 (NIH)
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Human Immunodeficiency Virus; HIV
Keywords: transition of care; adolescent
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Methods; Telemedicine; Standard of Care

STUDY DESIGN:
Intervention Model Description: This study uses a stepped-wedge, delayed implementation randomized clinical trial design, to measure the effectiveness of the interventions compared to standard of care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- In-person adolescent-friendly service (iPAS) intervention: (Experimental): Adolescents at study clinics who score low or intermediate on transition readiness during screening will be invited to enroll in the study. Adolescents attending clinics randomized to the in-person supported adolescent friendly services will attend their clinic after school hours on a designated day or on weekends dedicated for adolescent care monthly for 9 months.
  Interventions: Behavioral: In-person adolescent-friendly service (iPAS) intervention
- mHealth (InTSHA) intervention (Experimental): Adolescents at study clinics who score low or intermediate on transition readiness during screening will be invited to enroll in the study. Adolescents attending clinics randomized to the mHealth intervention will receive the InTSHA intervention based in the Got Transition elements and the SMART model for 9 months.
  Interventions: Behavioral: mHealth (InTSHA) intervention
- Standard of Care/Delayed Intervention (Active Comparator): Adolescents at study clinics who score low or intermediate on transition readiness during screening will be invited to enroll in the study. Adolescents attending clinics randomized to deliver the standard of care before transitioning to adult care in their standard local adult clinic. Participants will be invited to receive the intervention the clinic is randomized to deliver when the 9 month period of administering the standard of care is complete.
  Interventions: Behavioral: Standard of Care
- Healthcare Providers (No Intervention): Healthcare providers working at one of study clinics, administering the study intervention selected for that clinic.
- Observational cohort (No Intervention): Adolescents at study clinics who score high on transition readiness during screening will not be invited to enroll in the study but will be asked for their consent to have their clinic records reviewed for medical records, retention data and transition readiness data. They will also complete a questionnaire at Months 9, 18, and 24.

INTERVENTIONS:
Behavioral: In-person adolescent-friendly service (iPAS) intervention — Monthly visits take place in a group setting with sessions led by peer educators. Clinical staff and peer educators are trained in care of adolescents using the Right to Care training materials. During their clinic visit, adolescents are evaluated individually by a healthcare provider and receive their supply of ART. In addition, adolescents participate in scheduled group team-building activities including dancing, sports, music and receive group counseling facilitated by peer educators. Nine group counseling sessions will discuss the topics of: HIV disclosure, alcohol and substance abuse, HIV knowledge, ART adherence and HIV resistance, goal setting and career planning, sexual and reproductive health, HIV stigma, healthcare navigation and self-advocacy, and healthy relationships. The half-day sessions will end with the provision of a meal. After completion of the 9-month intervention, adolescents will transition to adult care in their standard local adult clinic.
  Arms: In-person adolescent-friendly service (iPAS) intervention:
Behavioral: mHealth (InTSHA) intervention — The InTSHA intervention is based on Got Transition elements (two-way messaging between adolescents and healthcare providers) and the SMART model. The SMART model focuses on modifiable factors of transition preparation through content delivery, facilitated discussions, online meet ups and consultation with the healthcare team. The intervention consists of 9 modules delivered monthly by group chat. The topics of the modules are: HIV disclosure, alcohol and substance abuse, HIV knowledge, ART adherence and HIV resistance, goal setting and career planning, sexual and reproductive health, HIV stigma, healthcare navigation and self-advocacy, and healthy relationships. Outside of scheduled group chat sessions, adolescents have access to the chat group to check in with members, review content of the sessions, or to comment or ask additional questions. After completion of the 9-month intervention, adolescents will transition to adult care in their standard local adult clinic.
  Arms: mHealth (InTSHA) intervention
Behavioral: Standard of Care — Adolescents in standard of care are seen every three months by clinicians and collect medication monthly at an on-site pharmacy during regular weekdays. Individual counseling delivered by counselors or social workers is available when necessary. Staff at all clinics receive training in adolescent-friendly services (AFS) through the Right to Care training materials.
  Arms: Standard of Care/Delayed Intervention

SUMMARY:
This is a cluster randomized controlled trial determining the effectiveness of in-person or mHealth-based adolescent-friendly transition interventions compared to standard care on retention in care and viral suppression among adolescents living with HIV who have low transition readiness. Participants are adolescents living with HIV ages 15 to 19 years old in KwaZulu-Natal, South Africa.

DETAILED DESCRIPTION:
South Africa has the highest number of adolescents living with HIV in the world, yet adolescents are poorly prepared for transition from pediatric to adult services. For a large majority of South Africans living with HIV, antiretroviral therapy (ART) was not available until 2004. This delay contributed to nearly 500,000 perinatal HIV infections in the late 1990s and early 2000s. With large scale-up efforts and improved access to ART in recent years, survivors of perinatal HIV infection are now reaching adolescence and beyond. As the wave of adolescents living with perinatally-acquired HIV matures, an estimated 320,000 adolescents will transfer from pediatric- or adolescent-based clinics to adult services in the next 10 years in South Africa. Although the mother-to-child HIV transmission rates in South Africa have decreased to less than 2%, thousands of infants are still being born with HIV each year ensuring that adolescent HIV will be an issue for many years. Currently, adolescents living with perinatally-acquired HIV enter adult care at variable ages and developmental stages, typically without necessary preparation or support through the process.

The transition from pediatric to adult services for adolescents living with HIV is a critically vulnerable time during which there is a high risk for disengagement from care and resultant morbidity and mortality. Despite an overall decrease in global HIV-related mortality, HIV remains the leading cause of death among adolescents living in South Africa where less than 50% of adolescents living with HIV are virally suppressed. Globally, disruptions related to transitioning from pediatric to adult care have been associated with high rates of HIV drug resistance, virologic failure, progression to AIDS and mortality. In South Africa, older adolescents (>15 years old) had lower viral suppression rates than younger adolescents at the time of transfer to general clinics.

Studies of in-person adolescent support groups (teen/adherence clubs) and adolescent-friendly services have shown mixed results in mitigating the poor outcomes of adolescents living with HIV. In-person adherence clubs have improved long-term adherence to ART among adults. However, the adherence or teen club models among adolescents living with HIV have shown mixed results.

The delivery of healthcare through portable mobile devices (mHealth) interventions have potential to remedy the challenges along the HIV continuum of care faced by adolescents living with HIV but larger, adequately powered randomized trials are needed. Adolescents in South Africa commonly communicate via social media to gain social support and health information from their peers and the use of social media for health expanded during the coronavirus infection 2019 (COVID-19) pandemic. mHealth strategies thus provides the opportunity to reach adolescents regularly using a preferred format, which could be utilized to improve the reach and impact of adolescent-focused interventions.

The Social-ecological Model of Adolescent and Young Adult Readiness to Transition (SMART) highlights modifiable targets of intervention that can improve transition care for adolescents living with HIV. The SMART model incorporates modifiable factors such as knowledge, skills/self-efficacy, relationships, and social support that can be targets of interventions to improve transition care. Medical care during adolescence is typically complicated by increased risk-taking behavior, as well as decreased caregiver involvement, which occur during a time of rapid physical, emotional, and cognitive development. When adolescents transition to adult care, they often do not receive the coordinated services that they received under pediatric care. The SMART model emphasizes eight modifiable factors, three key stakeholders (adolescents, caregivers, and clinicians) and their interconnected relationship in influencing successful transition to adult care. Using the SMART model, interventions delivered in-person or virtually can address the modifiable factors in the model to improve transition care for adolescents living with HIV but rigorous clinical trials are needed to prove effectiveness.

The researchers have developed and validated the first transition readiness assessment for adolescents living with HIV in South Africa and demonstrated its utility in predicting viral suppression in adult care. Through the development and validation of the HIV Adolescent Readiness to Transition Scale (HARTS) the researchers found that higher ratings reflecting HIV disclosure, healthcare navigation, self-advocacy, and health literacy were predictive of viral suppression after transition to adult care for adolescents living with HIV in South Africa. Using the HARTS in addition to demographic data associated with viral suppression after transition to adult care, the researchers created a transition readiness score to assist clinicians in determining which adolescents may benefit from additional services prior to transitioning to adult care.

Clinics in KwaZulu-Natal, South Africa are randomized to deliver an in-person adolescent-friendly service (iPAS) intervention, mHealth InTSHA intervention, or standard of care to adolescents receiving care at those clinics who score low or intermediate when screened for transition readiness. After the first 9 months of the study, the clinics randomized to deliver standard of care will begin delivering either the iPAS or InTSHA interventions for the next 9 month period. Adolescents participate in the intervention occurring at the clinic they attend for 9 months and complete surveys at baseline, after the 9 month intervention, and a final survey at the end of the study (15 or 24 months after enrollment). Adolescents with high scores when screened for transition readiness will comprise an observational cohort where data will be abstracted from medical records and they will complete questionnaires at 9, 18, and 24 months.

ELIGIBILITY:
Inclusion Criteria for Adolescent Participants:

* Aged 15 to 19 years at enrollment
* Living with perinatally-acquired HIV
* Receiving ART for at least 6 months
* Aware of their HIV status
* Scoring low to intermediate on transition readiness assessment (intervention cohort only)

Inclusion Criteria for Healthcare Providers:

* Profession as a healthcare provider
* Working at one of the designated clinics
* Involvement with adolescents before, during or after transition to adult care

Exclusion Criteria for all participants:

* Inability to read and/or speak English or Zulu
* Severe mental or physical illness preventing participation in informed consent activities
* Anticipated move out of clinic area in the next 12 months

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-02-02 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Retained in Care | After the 9 month intervention (Month 9 or Month 18)
  Clinic patients are considered to be retained in care if 80% of ART pharmacy refills are filled on time (< 7days from scheduled date) and 80% of scheduled clinic appointments are attended.
Change in Number of Participants with Viral Suppression | Baseline, After the 9 month intervention (Month 9 or Month 18)
  HIV-1 viral load is measured in viral copies per milliliter (mL) of blood and viral suppression is defined as <200 copies/ml.

SECONDARY OUTCOMES:
Acceptability of Intervention Measure (AIM) Score | Baseline, After the 9 month intervention (Month 9 or Month 18)
  Acceptability of the intervention is assessed with the AIM questionnaire. The AIM questionnaire has 4 items asking respondents how much they agree with statements such as "the intervention is appealing to me". Responses are given on a 5-point scale where "completely disagree" = 1 and "completely agree" = 5. Total scores range from 4 to 20 where higher scores indicate greater feelings of acceptability.
Intervention Appropriateness Measure (IAM) Score | Baseline, After the 9 month intervention (Month 9 or Month 18)
  Appropriateness of the intervention is assessed with the IAM questionnaire. The IAM questionnaire has 4 items asking respondents how much they agree with statements such as "the intervention seems applicable". Responses are given on a 5-point scale where "completely disagree" = 1 and "completely agree" = 5. Total scores range from 4 to 20 where higher scores indicate greater feelings that the intervention is appropriate.
Feasibility of Intervention Measure (FIM) Score | Baseline, After the 9 month intervention (Month 9 or Month 18)
  Feasibility of the intervention is assessed with the FIM questionnaire. The FIM questionnaire has 4 items asking respondents how much they agree with statements such as "the intervention seems possible". Responses are given on a 5-point scale where "completely disagree" = 1 and "completely agree" = 5. Total scores range from 4 to 20 where higher scores indicate greater feelings that the intervention is feasible.
HIV Adolescent Readiness for Transition Scale (HARTS) Score | Baseline, Month 9, Month 18, Month 24
  The HIV Adolescent Readiness for Transition Scale (HARTS) includes 16 items that are responded to on a 5-point scale where 0 = no, 1 = no, but I am learning, 2 = yes, a little bit, 3 = yes, almost always, and 4 = yes, always. Total scores range from 0 to 64 and higher scores indicate greater readiness to transition to adult care.
Participation Rate | Baseline, After the 9 month intervention (Month 9 or Month 18)
  Adoption of the intervention is examined as the number of adolescent patients enrolling in the study. Adoption of the intervention is considered successful with a participation rate threshold of >70%.
Intervention Fidelity | Up to Month 24
  Healthcare providers will complete an intervention checklist monthly during the intervention. A threshold of >80% of intervention checklist items is considered to be fidelity to the intervention.
Cost of the Intervention | After the 9 month intervention (Month 9 or Month 18)
  Cost of the intervention is assessed through time and motions studies. Time and motion studies involve counting the time a healthcare provider takes to prepare and deliver the intervention and how long (in hours) each session takes.
Intervention Completion Rate | After the 9 month intervention (Month 9 or Month 18)
  Completion of the intervention is examined as the number of adolescent participants who complete the study.
Percent of Clinic Visits Attended | Month 18, Month 24
  Sustained effectiveness of the study is examined as the percentage of scheduled clinic appointments that are attended, post-transitioning to care through an adult clinic. Attending at least 80% of scheduled clinic appointments is considered successful retention-in-care.
Percent of On Time Pharmacy Refills | Month 18, Month 24
  Sustained effectiveness of the study is examined as the percentage of ART pharmacy refills that are filled within 7 days from the scheduled date, post-transitioning to care through an adult clinic. Refilling at least 80% of ART pharmacy on time (< 7 days past the scheduled date) is considered successful retention-in-care in terms of pharmacy refills.

OTHER OUTCOMES:
Child and Adolescent Social Support Scale (CASSS) Score | Baseline, After the 9 month intervention (Month 9 or Month 18)
  Social support from peers is assessed using 10 items of the Child and Adolescent Social Support Scale (friend support subscale). Responses are given on a 6-point scale where 1 = never and 6 = always. Total scores range from 10 to 60, where higher scores represent greater social support from peers.
Rosenberg's Self-Esteem Scale Score | Baseline, After the 9 month intervention (Month 9 or Month 18)
  The Rosenberg's Self-Esteem Scale is a 10-item instrument assessing self-esteem. Responses are given on a 4-point scale where 0 = strongly disagree and 3 = strongly agree. Total scores range 0 to 30 and higher scores indicate greater self-esteem.
Patient Health Questionnaire (PHQ-9) Score | Baseline, After the 9 month intervention (Month 9 or Month 18)
  The PHQ-9 is a 9-item self-report questionnaire developed to identify patients at risk for depression. Participants report how often they have been bothered by specific symptoms of depression on a scale of 0 (not at all) to 3 (nearly every day). Higher scores indicate greater symptoms of depression. A score of ≥ 9 indicates clinically significant symptoms.
Internalized AIDS-Related Stigma Scale (IA-RSS) Score | Baseline, After the 9 month intervention (Month 9 or Month 18)
  The IA-RSS assesses several dimensions of stigma concerning HIV status. The instrument includes 6 items adapted form the AIDS-Related Stigma scale. Statements about hesitancy to disclose HIV status and feelings of shame are responded to as 0 = Disagree and 1 = Agree. Total scores range from 0 to 6 with higher scores indicating increased internalized stigma.
Working Alliance Inventory (WAI) Score | Baseline, After the 9 month intervention (Month 9 or Month 18)
  A modified version of the Working Alliance Inventory is used to measure how connected participants feel to the clinical staff and medical team. Ten items are responded to on a 4-point scale where 0 = strongly disagree and 3 = strongly agree. Total scores range from 0 to 30 where higher scores indicate increased feelings of connection with clinical staff.

CONTACTS AND LOCATIONS:
Overall Officials: Brian C Zanoni, MD, MPH, Principal Investigator — Emory University; Mohendran Archary, MBchB, Principal Investigator — King Edward VIII Hospital
Locations (1):
- King Edward VIII Hospital, KwaKhangela, South Africa

IPD SHARING:
Plan to Share IPD: Yes
De-identified, individual participant data will be made available for sharing, including demographic information, clinic information, and study and survey data.
Supporting Information: Study Protocol
Time Frame: Data will be made available for sharing following publication of results from this study.
Access Criteria: Data will be made available for sharing through the Emory Dataverse. The Dataverse website can be accessed by any researcher for secondary analyses.